CLINICAL TRIAL: NCT07302828
Title: Effect of Double Nutri® Liposomal Encapsulation Technology on Human Absorption of Vitamin C and Glutathione Liquid Sachet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25-098-A
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Vitamin C; Glutathione
Keywords: vitamin c; glutathione; liposomal; human bioavailability; Double Nutri
MeSH Terms: interventions — Ascorbic Acid; Glutathione; Liposomes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C and Glutathione without liposome (Active Comparator): Each administration consists of two sachets, with each sachet containing 1,000 mg of vitamin C and 60 mg of glutathione
  Interventions: Dietary Supplement: Vitamin C and Glutathione without liposome
- Liposomal Vitamin C and Glutathione (Experimental): Each administration consists of two sachets, with each sachet containing 1,000 mg of vitamin C and 60 mg of glutathione, and the test sample is processed using the Double Nutri liposomal technology
  Interventions: Dietary Supplement: Liposomal Vitamin C and Glutathione

INTERVENTIONS:
Dietary Supplement: Vitamin C and Glutathione without liposome — Each administration consists of two sachets, with each sachet containing 1,000 mg of vitamin C and 60 mg of glutathione.
  Arms: Vitamin C and Glutathione without liposome
Dietary Supplement: Liposomal Vitamin C and Glutathione — Each administration consists of two sachets, with each sachet containing 1,000 mg of vitamin C and 60 mg of glutathione, and the product is processed using the Double Nutri liposomal technology.
  Other Names: GLUTA BRIGHT; Double Nutri Vitamin C and Glutathione
  Arms: Liposomal Vitamin C and Glutathione

SUMMARY:
The objective of this study is to evaluate whether Double Nutri® liposomal encapsulation technology can enhance the oral absorption of liquid vitamin C and glutathione supplements in humans.

DETAILED DESCRIPTION:
This study is a single-center, self-controlled crossover human trial designed to evaluate the differences in blood concentration changes and bioavailability following a single oral dose of liquid vitamin C and glutathione supplements.

Healthy adult participants aged 18 years and older will be enrolled. Each participant will complete two study sessions, with a minimum washout period of 7 days between sessions. On each study day, venous blood samples will be collected prior to test product administration (0 minutes) to assess vitamin C levels, glutathione levels, complete blood count, blood lipids, blood glucose, and liver and kidney function indicators.

After baseline blood collection, a standardized breakfast will be provided and consumed within 10 minutes, followed by administration of the test product. Venous blood samples will then be collected at 0.5, 1, 2, 4, 6, and 8 hours post-intake to measure vitamin C and glutathione concentrations. Lunch will be provided after the 4-hour blood draw, and dinner will be provided after the 8-hour blood draw. Identical meals will be provided during both study sessions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older, of any sex, who are willing to sign the informed consent form and are able to fully comply with all study procedures.

Exclusion Criteria:

* Pregnant or breastfeeding women, or individuals unwilling to use physical contraceptive methods during the study period, such as condoms or intrauterine devices (IUDs).
* Employees of TCI Co., Ltd and their family members.
* Individuals who, within 30 days prior to study initiation, have been taking vitamin C supplements at doses greater than 200 mg per day, glutathione supplements at doses greater than 100 mg per day, or medications that may affect endogenous vitamin C or glutathione levels, such as oral contraceptives and estrogen preparations (including ethinylestradiol, desogestrel, gestodene, drospirenone, cyproterone acetate), or acetaminophen.
* Individuals with chronic gastrointestinal diseases (including irritable bowel syndrome [IBS], inflammatory bowel disease [IBD], chronic diarrhea, Crohn's disease, celiac disease, bowel control disorders/fecal incontinence, pancreatitis, peptic ulcer disease, colorectal cancer, short bowel syndrome, and ulcerative colitis), a history of epilepsy or seizures, liver or kidney disease, malignancy, endocrine disorders, psychiatric disorders, alcohol or drug abuse, or other significant organic diseases based on medical history.
* Individuals who have undergone gastrointestinal surgery, organ transplantation, or other major surgical procedures.
* Individuals who experienced acute gastroenteritis within two weeks prior to study initiation.
* Individuals with a known allergy to any components of the testing samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Blood vitamin C level (ug/mL) | at 8 hours after taking test sample
  Blood vitamin C levels will be measured at fasting and at 0.5, 1, 2, 4, 6, and 8 hours post-intake.
Blood glutathione level (μmol/L) | at 8 hours after taking test sample
  Whole blood glutathione levels will be measured at fasting and at 0.5, 1, 2, 4, 6, and 8 hours post-intake.

CONTACTS AND LOCATIONS:
Overall Officials: Tong-Lin Wu, Principal Investigator — TCI Co., Ltd.
Locations (1):
- TCI Co., Ltd, Taipei, Taiwan